CLINICAL TRIAL: NCT05851924
Title: Total Neoadjuvant NALIRIFOX Plus Ablative Dose Radiation Therapy for Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma
Brief Title: A Study of NALIRIFOX in Combination With Radiation Therapy in People With Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ipsen (Industry); Pancreatic Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-027
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: NALIRIFOX; Ablative Dose Radiation; 23-027
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NALIRIFOX + AD-XRT and capecitabine (Experimental): Patients will receive neoadjuvant chemotherapy for 4 months. Patients will undergo a CT scan at 8 weeks and 16 weeks after the start of neoadjuvant chemotherapy to assess treatment response. Patients without disease progression will then undergo AD-XRT for 15 to 25 fractions (3 to 5 weeks). Patient's whose disease is deemed resectable based on their re-evaluating imaging, will be recommended surgical intervention with consideration for laparotomy or laparoscopy if deemed appropriate at multidiscplinary cancer conference review.
  Interventions: Drug: NALIRIFOX; Combination Product: AD-XRT and Capecitabine

INTERVENTIONS:
Drug: NALIRIFOX — Patients will receive NALIRIFOX for a total of 4 months. NALIRIFOX will be administered on days 1 and 15 of a 4-week cycle for 4 cycles until completion of therapy, intolerable toxicity, or until the development of criteria for removal from the study.
  Liposomal irinotecan: 50 mg/m2 IV over the course of 90 minutes (±10 minutes) on days 1 and 15 of every 4-week cycle.
  Oxaliplatin: 60 mg/m2 IV over the course of 120 minutes (±10 minutes) on days 1 and 15 of every 4-week cycle.
  Leucovorin: 400 mg/m2 IV over the course of 30 minutes (±5 minutes) on days 1 and 15 of every 4-week cycle.
  5-FU: 2400 mg/m2 IV over the course of 48 hours (or until the infusion is complete) on days 1 and 15 of every 4-week cycle
Combination Product: AD-XRT and Capecitabine — The interval between completion of induction chemotherapy and initiation of AD-XRT will be 2-6 weeks. The patient will be concurrently treated with capecitabine (1000-1500 mg flat BID PO Monday to Friday) with radiation, as per standard dosing regimens at MSK.

SUMMARY:
The researchers are doing this study to find out whether using the chemotherapy regimen NALIRIFOX in combination with ablative dose radiation therapy (AD-XRT) and the standard chemotherapy drug capecitabine is an effective treatment approach for people with locally advanced or borderline resectable pancreatic ductal adenocarcinoma (PDAC) before surgery. This type of treatment approach is called total neoadjuvant therapy (TNT). The researchers will also look at whether the sequence of the treatment approach (NALIRIFOX + ADXRT and capecitabine followed by surgery, when it is possible) is effective and causes few or mild side effects in participants. An important purpose of the study is to see how the study treatment (NALIRIFOX + AD-XRT and capecitabine) affects participants' quality of life. The researchers will measure quality of life by having participants fill out questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been informed about the nature of the study, has agreed to participate in the study, and has signed the informed consent form before participation in any study-related activities.
2. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.

   Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, DCIS, stage I prostate cancer, and basal cell or squamous cell carcinoma of the skin.
3. A multidisciplinary discussion has been undertaken/planned which can include (a) discussion with medical/surgery oncology, (b) Hepatopancreaticobiliary Disease Management Team conference presentation, (c) direct consultation, with confirmation on consensus plan for TNT strategy and potential for future surgery. This plan needs to be documented in the medical record prior to initiation of treatment.
4. Male or nonpregnant and nonlactating female aged ≥18 years.

   1. Women of child-bearing potential (i.e., fertile, following menarche, and until becoming postmenopausal unless permanently sterile; permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) must test negative for pregnancy at the time of screening on the basis of a urine or serum pregnancy test. Postmenopausal women are defined as those who have had an absence of menstruation for at least 2 years. If necessary, follicle-stimulating hormone results >50 IU/L at screening are confirmatory in the absence of a clear postmenopausal history.
   2. Female subjects of reproductive potential must agree to use two effective methods of birth control during the study and for 9 months after the last dose of study medication.
   3. Male subjects must agree to use condoms during the study and for 4 months after the last dose of study medication'

Disease-specific inclusion criteria:

1. Histologically or cytologically confirmed PDAC that has not been previously treated.
2. Radiographically BR or LA PDAC in accordance with the NCCN 2.2021 definition, without evidence of distant metastases by CT.
3. Inoperable status after surgical exploration due to presence of locally advanced, unresectable disease without metastases, in patients who have recovered from surgery, is allowed.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Hematological, biochemical, and organ function inclusion criteria:

   1. Absolute neutrophil count (ANC) ≥1500/mm^3 without the use of hemopoietic growth factors within 7 days before treatment
   2. Platelet count ≥100,000/mm^3 .
   3. International normalized ratio (INR) <1.5 unless the patient is receiving anticoagulation therapy, in which case a therapeutic INR is acceptable. Anticoagulation therapy with low-molecularweight heparin or warfarin, whether medically indicated, is permitted.
   4. Adequate renal function, as evidenced by serum/plasma creatinine level <1.6 mg/dL

Exclusion Criteria:

1. Presence of metastatic pancreatic cancer (M1 disease)
2. Any other medical or social condition deemed by the investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, and participate in the study or who is likely to interfere with the interpretation of the results.
3. Unwilling or unable to comply with study procedures and/or study visits.
4. Medical co-morbidities, that preclude major abdominal surgery
5. Histologic diagnosis other than adenocarcinoma; however, adenosquamous variants are acceptable.
6. Receipt of chemotherapy, prior abdominal radiotherapy, and/or definitive resection for pancreatic cancer.
7. Grade >2 neuropathy.
8. Pregnant and/or nursing.
9. Uncontrolled active infection, which would preclude with the exception of resolving cholangitis which in the investigator opinion would render the treatment hazardous.
10. Known hypersensitivity to any of the components of the chemotherapeutic agents
11. Receipt of concurrent investigational therapy or within 30 days of protocol initiation.

    Additional criterion for the immunoPET imaging sub-study (n=20)
12. Previous anaphylactic reaction to human, humanized or chimeric antibody.
13. Refusal or inability to tolerate the scanning procedure (e.g. due to claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
event-free survival (EFS) | up to 16 weeks
  events defined as: 1) progression [local or systemic progression, per RECIST], 2) recurrence [recurrent disease following resection], or 3) death due to any cause

SECONDARY OUTCOMES:
overall survival (OS) rate | up to 5 years
  defined as the time from enrollment to death from any cause. Patients alive are censored at the date of last contact

CONTACTS AND LOCATIONS:
Overall Officials: Alice Wei, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm